CLINICAL TRIAL: NCT05038839
Title: A Phase I Study of Cabozantinib and Pamiparib to Evaluate Triple Inhibition of PARP, VEGFR and c-MET in Advanced Homologous Recombination Deficient Malignancies
Brief Title: Cabozantinib and Pamiparib for the Treatment of Advanced of Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0308; NCI-2021-03248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0308 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-18; First posted 2021-09-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: interventions — cabozantinib; pamiparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib, pamiparib) (Experimental): Patients receive cabozantinib PO QD and pamiparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Drug: Pamiparib

INTERVENTIONS:
Drug: Cabozantinib — Given PO
Drug: Pamiparib — Given PO
  Other Names: BGB-290; PARP Inhibitor BGB-290

SUMMARY:
This phase I trial finds the best dose and side effects of cabozantinib and pamiparib in treating patients with solid tumors that have spread to other places in the body (advanced) or does not respond to treatment (refractory). Cabozantinib and pamiparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) or maximum administered dose (MAD) and dose-limiting toxic effects (DLTs) of cabozantinib and pamiparib.

II. To define the safety profiles of cabozantinib and pamiparib.

SECONDARY OBJECTIVES:

I. To perform plasma pharmacokinetic analyses of cabozantinib and pamiparib interaction.

II. To evaluate patient reported outcomes (PRO). III. To evaluate pre-identified mutations in circulating free deoxyribonucleic acid (DNA) (cfDNA) by next generation sequencing (NGS).

IV. To estimate complete responses (CRs), partial responses (PRs), stable disease >= 6 months (SD >= 6months), progression free survival (PFS) and overall survival (OS).

V. To relate changes in phosphorylated AKT (pAKT), phosphorylated ERK2 (pERK2), phosphorylated c-MET (pc-MET), phosphorylated PARP1 (PARP1-pY907), phosphorylated histone H2A variant H2AX (gamma-H2AX) and RAD51 in tumor specimens with antitumor efficacy.

VI. To relate cancer-associated mutations at baseline with antitumor efficacy. VII. To explore potential biomarkers of acquired resistance by comparing molecular signatures at baseline with those at time of relapse in patients in whom SD >= 6 months/CR/PR or a mixed response are documented, by next-generation deep sequencing or more sophisticated techniques.

OUTLINE: This is a dose-escalation study.

Patients receive cabozantinib orally (PO) once daily (QD) and pamiparib PO twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced solid tumors refractory to standard-of-care (SOC) therapy; or no SOC therapy; or declined SOC. During dose expansion, patients have to have one of the following genetic and pathologic features as defined in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory as well:

  * A deleterious BRCA1 or BRCA2 mutation (germline or somatic)
  * A surrogate biomarker for HRD: deleterious mutation or deletion of MRE11, RAD50, NBS1, ATM, ATR, CHEK1, CHEK2, PALB2, ARID1A, Fanconi anemia genes, and PTEN, or loss of PTEN by IHC, amplification of EMSY, etc
* Patients in the dose-escalation phase must have evaluable and/or measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Patients in the dose expansion phase must have measurable disease per RECIST 1.1 and at least one additional lesion that can be biopsied
* Patients age >= 18 years
* For women of child-bearing potential (women who have not been postmenopausal for at least one year or are not surgically sterile) and all men, agreement to use highly effective contraception (e.g., hormonal contraception, barrier device, or abstinence) prior to study entry for the duration of study participation and for 180 days after the last dose of the study agents. Nonsterile males must avoid sperm donation for the duration of the study and for at least 6 months after the last dose of the study agents
* White blood cell count >= 2,500/uL, without granulocyte colony-stimulating factor support (within 14 days before first dose of study treatment)
* Absolute neutrophil count (ANC) >= 1,500/uL, without granulocyte colony-stimulating factor support (within 14 days before first dose of study treatment)
* Hemoglobin >= 9 g/dL (within 14 days before first dose of study treatment)
* Platelets >= 100,000/uL, without transfusion (within 14 days before first dose of study treatment)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (upper limit of normal), or total bilirubin < 3.0 x ULN with direct bilirubin =< ULN in patients with well documented Gilbert's syndrome (within 14 days before first dose of study treatment)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (AKP) =< 3 x ULN. AKP =< 5 x ULN with documented bone metastases (within 14 days before first dose of study treatment)
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance >= 45 mL/min by the Cockcroft-Gault method (within 14 days before first dose of study treatment)
* Serum albumin >= 2.8 g/dL (within 14 days before first dose of study treatment)
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg (=< 113.2 mg/mmol), or 24-h urine protein =< 1 g (within 14 days before first dose of study treatment)
* Prothrombin time (PT)/institutional normalized ratio (INR) or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN if not on therapeutic anticoagulation (within 14 days before first dose of study treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Ability to read and fully understand the requirements of the trial, willingness to comply with all trial visits and assessments, and willingness and ability to sign an Institutional Review Board (IRB)-approved written informed consent document
* No palliative radiation therapy delivered to the sole target lesions immediately before or during the study
* Ability to take oral medications without medical history of malabsorption or other chronic gastrointestinal disease, or other conditions that may hamper compliance and/or absorption of the study agents
* No prior treatment with simultaneous inhibition of PARP and VEGF with or without c-MET inhibition (patients may have prior therapy targeting only the c-MET, VEGF, or PARP pathway). However, prior treatment with cabozantinib is not allowed
* Willing to provide an archival tissue block, or 10 formalin-fixed paraffin-embedded (FFPE) slides

Exclusion Criteria:

* Any treatment specifically for systemic tumor control given within 3 weeks before the initiation of the study drugs, within 2 weeks if cytotoxic agents were given weekly, within 4 weeks if cytotoxic agents were given once every 3 to 4 weeks, within 6 weeks for nitrosoureas or mitomycin C, within 5 half-lives for targeted agents with half-lives and pharmacodynamic effects lasting < 5 days (a minimum of 10 days is required), or failure to recover from toxic effects of any therapy before the initiation of the study drugs
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Major surgery (e.g., laparoscopic nephrectomy, gastrointestinal (GI) surgery, removal or biopsy of brain metastasis) within 4 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Unresolved grade 1 or higher toxicity from prior therapy that is clinically significant
* Patient has an inability to swallow oral medications. Note: Patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN)
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.

      * Note: Subjects with a diagnosis of incidental, subsegmental pulmonary embolism (PE) or deep vein thrombosis (DVT) within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment.
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.

      * Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
  * Other clinically significant disorders that would preclude safe study participation.

    * Serious non-healing wound/ulcer/bone fracture.
    * Uncompensated/symptomatic hypothyroidism.
    * Moderate to severe hepatic impairment (Child-Pugh B or C)
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment
* No other anticancer-therapy (chemotherapy, immunotherapy, hormonal anti-cancer therapy, radiotherapy [except for palliative local radiotherapy]), biological therapy or other novel agent is to be permitted while the patient is receiving study medication. Patients on LHRH analogue treatment for more than 6 months are allowed entry into the study and may continue at the discretion of the Investigator
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment. Leptomeningeal or lymphangitic carcinomatosis is not allowed
* Patient has had prescription or non-prescription drugs or other products known to be moderate to strong inhibitors or inducers of CYP3A which cannot be discontinued at least 5 half-lives if known, or 14 days if unknown prior to day 1 of dosing, and withheld throughout the study until 2 weeks after the last dose of study drug
* Herbal preparations are not allowed throughout the study. These herbal medications include but are not limited to: St. John's wort, kava, ephedra (ma hung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng. Patients should stop using these herbal medications 5 half-lives if known or 14 days if unknown prior to first dose of study treatment
* Any known hypersensitivity or contraindication to the components of the study drugs
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment [QTcf = QT/(RR^0.33); RR interval = 60/heart rate], or congenital long QT syndrome.

  * Note: If a single electrocardiography (ECG) shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility
* Pregnant or breastfeeding women
* Serious active infection at the time of study entry, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Grade 2 or higher peripheral neuropathy
* Human immunodeficiency virus requiring highly active antiretroviral therapy (HAART) treatment due to unknown drug-drug interactions or has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or C virus (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [quantitative] is detected) infection: patients who have had active hepatitis B virus [HBV] or HCV infections in the past but have evidence of viral clearance as shown by negative viral load, i.e., undetectable HBV DNA or HCV RNA, will be eligible
* Lesions invading or encasing any major blood vessels. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Vaccination with live vaccine within 4 weeks of treatment start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Descriptive statistics will be provided on the grade and type of toxicity by dose level.
Dose-limiting toxicities | Up to 28 days
Recommended phase 2 dosage | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org